CLINICAL TRIAL: NCT00916565
Title: The Evaluation of Cow Milk-Based Formulas - Functional Proteins
Brief Title: Evaluation of Cow Milk-Based Formulas - Functional Proteins
Status: Completed | Type: Observational
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Bryan Liu, Mead Johnson Nutrition
Other Study IDs: 3378-3
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: optimize nutritional content of infant formula; Infant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Experimental milk-based infant formula
- Control milk-based infant formula
- Breastfed Reference Group

SUMMARY:
The purpose of this study is to look at the function of infant formula components to optimize the nutritional content and functionality of a marketed routine infant formula.

ELIGIBILITY:
Inclusion Criteria:

* 10-18 days of age
* 37-42 weeks gestation
* birth weight 2500 g or more
* consuming one source of nutrition

Exclusion Criteria:

* metabolic or chronic disease
* acute infection
* feeding difficulties
* consumed complementary foods or donor milk
* steroid use

Ages: 10 Days to 18 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: formula-fed and breastfed infants
Sampling Method: Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2009-07

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Dr. Claude Ashley, Birmingham, Alabama
  - William Johnston, MD, Birmingham, Alabama
  - Lori Montgomery, MD, Little Rock, Arkansas
  - Edward Zissman, MD, Lake Mary, Florida
  - Harold Deulofeut MD, Plantation, Florida
  - Harold Deulofeut MD, Tamarac, Florida
  - Susan Carlson, Ph.D., Kansas City, Kansas
  - Joseph Leader, MD, Woburn, Massachusetts
  - Ann Grandjean, Ed. D, Omaha, Nebraska
  - Laurie Harris-Ford, MD, Clarksville, Tennessee
  - Beth Nauert, MD, Austin, Texas

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831